CLINICAL TRIAL: NCT03376906
Title: The Effects of High Intensity Interval Exercise With 1- and 3- Min Recovery Times in Obese
Brief Title: The Effects of High Intensity Interval Exercise in Obese
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Yokiny Silva, Physiotherapist, Federal University of Paraíba
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Interval exercise
Record Dates: First submitted 2017-02-20; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Obesity; Endothelial Dysfunction
Keywords: Obesity; aerobic exercise; interval exercise
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The subjects were welcomed for a visit to the Laboratory of Studies of Physical Training Applied to Health, where they performed an evaluation of body composition, maximal ergospirometric exercise test, and three experimental sessions in a random order, which were performed with a 96 h interval between them. In order to obtain the experimental session order, the researcher asked each subject to pick out random numbers that were inside an opaque envelope generated at www.randomizer.org.
  Before the experimental sessions, subjects were instructed to maintain a regular sleep pattern, and to not consume alcohol, caffeine or xanthines (coffee, chocolate, soft drinks and tea), take medication or exercise in the 24 h prior to the experimental protocol sessions. In addition, they were duly instructed to fill out the food registry (food recall).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obese Subjetcs (Experimental): The subjects were welcomed for a visit to the Laboratory of Studies of Physical Training Applied to Health, where they performed an evaluation of body composition, maximal ergospirometric exercise test, and three experimental sessions (HIIE 1, HIIE 3 and Control) in a random order, which were performed with a 96 h interval between them.
  Interventions: Procedure: HIIE 1; Procedure: HIIE 3; Procedure: Control

INTERVENTIONS:
Procedure: HIIE 1 — In the HIIE 1 session, all the subjects performed 10 stimuli of 1 min at high intensity (92% of VO2Max) with passive recovery (without exercise) of 1 min.
Procedure: HIIE 3 — In the HIIE 3 session, the subjects performed the same stimulus of the HIIE1, but with passive recovery of 3 min. Both protocols started with a warm-up of 5 min at 50% of the VO2Peak performed on a T2-100 GE Healthcare® treadmill (Lynn Medical, Wixon, Michigan, USA).
Procedure: Control — In the control session, participants remained seated for 30 min. During HIIE 1 and 2, HR and RPE were assessed immediately after stimulus intervals (ten measurements at each HIIE). In all sessions, the subjects remained in supine position to obtain hemodynamic measurements which were obtained before and at 10 min, 30 min and 60 min after the HIIE and control sessions.

SUMMARY:
Obesity is a complex and multifactorial disease. Excess weight is related to endothelial dysfunction, inflammation and oxidative stress which increases the risk for cardiovascular diseases. High-intensity interval exercise can release vasodilatory substances and promote increased muscle blood flow.

DETAILED DESCRIPTION:
This study evaluated the effects of the recovery interval duration (1 vs. 3 min) in high intensity interval exercise (HIIE) on the hemodinamics responses in obese individuals. Twelve obese subjects (27 ± 3.8 yrs) were evaluated, who underwent three experimental sessions with a randomized crossover design: one control session (no exercise) and two HIIE sessions with the same workload (10 x 1min @92%VO2max / 1[HIIE 1] or 3[HIIE 3] min @0%). Forearm blood flow (FBF) and blood pressure (BP) were measured before and after the experimental sessions. Heart rate and relative perceived exertion were assessed during HIIE.

ELIGIBILITY:
Inclusion criteria for the study were obesity and the conditions of being insufficiently active, non-smokers and without previous history of: heart disease, obstructive or restrictive pulmonary diseases, and orthopedic morbidities. Fifty-one (51) subjects were evaluated for eligibility, and 39 subjects were excluded after an initial interview since they did not meet the aforementioned inclusion criteria.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-06-05 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2017-01-30 (Actual)

PRIMARY OUTCOMES:
Forearm Blood Flow and Vascular Conductance | Up to 2 years
  Forearm muscular blood flow was obtained through the venous occlusion plethysmography technique (19). For this, a silicon tube filled with mercury and connected to a low-pressure transducer was placed around the forearm, 5 cm away from the humeral-radial joint, connected to a plethysmograph (Hokanson® / EC6 plethysmograph, Bellevue, Washington, USA). A cuff was placed around the wrist and another at the upper arm, and the wrist cuff was inflated to a supra-systolic level every 1 min before measurements start. The arm cuff was inflated above the venous pressure at 10 s intervals for a period of 7 to 8 s. The increase in tension in the silastic tube reflects the increase in the volume of the forearm, which indicates vasodilation. The muscle flow wave signal was collected and stored on the WINDAQ DI 200 DATAQ program. Vascular conductance in the forearm was calculated by the blood flow ratio in the forearm (mL.min-1.100mL-1) and mean arterial pressure (mmHg) multiplied by 100.

SECONDARY OUTCOMES:
Blood pressure | Up to 2 years
  Blood pressure values were obtained in a non-invasive manner, using an oscillometric method (Dixtal®, DX 2020; Manaus, Amazonas, Brazil). The occlusive cuff was positioned on the left ankle of the subject and was inflated minute by minute, providing systolic (SBP), diastolic (DBP) and mean (MBP) blood pressure values. For electrocardiogram (ECG) acquisition, three electrodes were placed on the thorax of the subjects in the bipolar position and DII derivation. After pre-amplification of the ECG signal, a conversion from analog to digital was performed, and later stored in a computer and processed by the WINDAQ DI-200 program (WinDaq DI-200, Akron, Ohio).
Heart rate | Up to 2 years
  Heart rate was monitored throughout the exercise session using a Polar RS800CX monitor (Polar®, Kempele, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Maria do Socorro B Santos, Ph.D., Study Director — Federal University of Paraíba

IPD SHARING:
Plan to Share IPD: No